CLINICAL TRIAL: NCT06414668
Title: ENERGY Expenditure of COmmuting to School
Brief Title: The ENERGYCO Study
Acronym: ENERGYCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); University of Jaén (Other); Navarra Institute for Health Research (Unknown); Centro de Investigación Biomédica en Red Fisiopatología de la Obesidad y Nutrición (Unknown); University of Otago (Other)
Responsible Party: Principal Investigator, Emilio Villa González, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENERGYCO
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Energy Expenditure; Physical Activity; Behavior; Body Composition
Keywords: Resting metabolic rate; Energy expenditure; Physical activity; Body composition; Cycling; School
MeSH Terms: conditions — Motor Activity; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycling group (Experimental): The intervention will include two Bikeability sessions and encouragements strategies will be carried out to complete the eight-weeks intervention based on cycling to and from school
  Interventions: Behavioral: Cycling Intervention Group
- Control group (No Intervention): The control group will keep their usual mode of commuting to and from school.

INTERVENTIONS:
Behavioral: Cycling Intervention Group — A eight-weeks school-based cycling program. The school-based cycling intervention consists of 2 Bikeability sessions of 60 min at Physical Education lessons in school, and will focus on promote biking through theory and practice lessons about cycle training skills including on-road training. In addition, participants will receive encouragement strategies, one for each week of the intervention, for cycling to and from school during eight weeks.
  Arms: Cycling group

SUMMARY:
The aims of this school-based cycling intervention called "ENERGY Commuting to school" (ENERGYCO) will be divided into two phases: Phase I will aim: 1) to design, test, and validate predictive equations for the objective quantification of the energy expenditure related to different modes of commuting to school (i.e., walking, cycling, motorized-vehicle); and 2) to quantify the energy expenditure of each mode of commuting to school using indirect calorimetry in adolescents; and Phase II will aim to evaluate the effect of a school-based cycling intervention on different health-related outcomes, such as energy expenditure, resting metabolic rate, basal metabolism, physical activity levels, body composition, muscle strength, cardiorespiratory fitness, blood pressure, physical literacy, motor competence, and psychosocial outcomes on Spanish adolescents.

DETAILED DESCRIPTION:
The ENERGYCO study is a cluster-randomized controlled trial focused on the energy expenditure associated with commuting to school. Phase I will aim to develop predictive equations for quantifying energy expenditure during different modes of commuting (walking, cycling, motorized-vehicle) and to measure energy expenditure using indirect calorimetry in adolescents. Phase II will assess the impact of a school-based cycling intervention on various health outcomes in Spanish adolescents, including energy expenditure, metabolic rate, physical activity levels, body composition, muscle strength, fitness, blood pressure, physical literacy, motor competence, and psychosocial outcomes. Phase I will involve recruiting approximately 50 adolescents to quantify energy expenditure during walking, cycling, and motorized-vehicle. For Phase II, a random sample of around 300 schoolchildren aged 12-16 from three Spanish cities will undergo a eight-week cycling intervention involving Bikeability sessions and encouragement strategies. Therefore, the ENERGYCO study aims to develop predictive equations for measuring energy expenditure during active commuting to school and assess the impact of a cycling intervention on adolescent health. It is expected to contribute significantly to research and society by providing insights into the effects of active commuting and cycling interventions on adolescent energy expenditure, physical and mental health.

ELIGIBILITY:
Inclusion Criteria:

1. the school has a specific space for parking bicycles and allows for their parking
2. the school does not have a specific school bus route
3. the school has at least two lines per class
4. at least eight students from the school will agree to participate in the study (i.e., presenting a signed parental consent).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of the resting metabolic rate | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of the resting metabolic rate using indirect calorimetry (Ominical)
Change of the daily energy expenditure | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of the energy expenditure using predictive equations developed during the Phase I of the stuy and validated against indirect calorimetry (Cosmed K5)

SECONDARY OUTCOMES:
Change of Physical activity levels | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of the physical activity levels using accelerometry and the "Youth Physical Activity Profile" questionnaire
Heart rate monitoring | During the 8 weeks when the participant will cycle to and from school
  Assessment of the intensity of the commuting by bike to and from school using a pulsometer
Resting heart rate monitoring | First weekend of the school-based cycling intervention
  Assessment of the resting heart rate using a pulsometer
Cycling skill assessment: Bikeability sessions | First week of the school-based cycling intervention
  Assessment of the cycling skills in a closed circuit
Change of physical fitness | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of cardiorespiratory fitness (Course Navette), muscular strength (analog dinamometer), and blood pressure (stethoscope )
Change of physical literacy | 8 weeks during both measurement points (Baseline and post-intervention)
  Assesment of phsychological, social, cognitive, and motor competence using the Spanish perceived physical literacy instrument for adolescents (PPLI-Q) and the Bruininks-Oseretsky Test of Motor Proficiency (BOT-2)
Change of anthropometric measures | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of height and weight, (e.g., weight and height will be combined to report BMI in kg/m^2)
Change of anthropometric measures | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of waist and neck circumference in centimeters
Change of body composition | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of fat free mass, fat mass, lean mass index, fat mass index, body fat percentage, visceral adipose tissue, and bone mineral content using Dual energy X-ray absorptimetry (DEXA)
Change of cognitive determinants | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of subjective norm, intention, perceived behavioral control and attitude using Questionnaire stages of change
Change of perceptions to active commuting to and from school | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of perceived barriers to active commute to school using the Barriers for active commuting to school questionnaire (BATACE)
Change in children's psychosocial variables | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of autonomy, competence, and relatedness using the Basic Pshychological Need Satisfaction Need in Active Commuting to and from School questionnaire (BPNS ACS)
Change in children's psychosocial variables | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of satisfaction and motivation to active commuting to and from school using the Behavioural Regulation in Active Commuting to and from School questionnaire
Change in children's psychosocial variables | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of self-Esteem and mental health using the Positive and Negative Affect Schedule and the Rosenberg Self-Esteem Scale (RSES)
Children sociodemographic characteristics | 8 weeks during both measurement points (Baseline and post-intervention)
  Participants self-report their age, school grade and class, gender, full postal address, bicycle owners through a student questionnaire
Parents sociodemographic characteristics | 8 weeks during both measurement points (Baseline and post-intervention)
  Parents self-report the school name, child name, age, gender, children´s gender, and full postal address, parental education level through a parents questionnaire
Family socioeconomic status | 8 weeks during both measurement points (Baseline and post-intervention)
  Children and parents self-report their family income using the Family Affluence Scale questionnaire (FAS III)
Change of parental perceptions | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of the parents´ barriers to allow their adolescent to active commuting to and from school using the Parental Perception of Barriers towards active commuting to school questionnaire (PABACS)
Distance home-school-home | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of the route characteristics using Google Maps and GPS
Weather | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of the Temperature (maximum, minimum, mean), total rainfall, and mean wind speed using data from the National Weather Data Bank
School characteristics | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of the school enrolment by electronic and manual search
School characteristics | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of the school socioeconomic status using Geographical Information System
School characteristics | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of the school engagement using data from the Ministry of Education and Vocational Training
City characteristics | 8 weeks during both measurement points (Baseline and post-intervention)
  Assessment of the population density and city income using data from the Tax Agency, Spanish Public Ministry of Finance and Public Administration of Spain

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided